CLINICAL TRIAL: NCT03554954
Title: Association Between Food/Nutrient Intake and Sleep Quality in Middle Aged and Older Population
Status: Completed | Type: Observational
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Jung Eun Kim, Assistant Professor, National University of Singapore
Other Study IDs: S1
Record Dates: First submitted 2018-04-22; First posted 2018-06-13 (Actual); Results first posted 2020-06-01 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Sleep
Keywords: Nutrients; Diet; Sleep Quality; Middle-aged adults; Older adults
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole Blood, Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sleep is essential to health. Quality of sleep, measure through indexes of sleep, is related to the incidence of obesity, type 2 diabetes, cardiovascular disease, hypertension, and premature death. Sleep pattern changes as people age. They tend to have a harder time falling asleep and more trouble staying asleep than when they were younger. Studies have shown that food/nutrient intake may be associated with sleep duration, quality, and patterns. Singapore's population is aging rapidly and improving their indexes of sleep may result in their health promotion.

DETAILED DESCRIPTION:
Sleep is essential to health and indexes of sleep including duration, quality, and patterning are related to the incidence of chronic diseases and premature death. Changes in sleep patterns are a part of the aging process and as people age, they tend to have a harder time falling asleep and more trouble staying asleep than when they were younger. Certain cross-sectional studies have shown that food/nutrient intake may be associated with sleep duration, quality, and patterns. In the last decade, Singapore's population has grown older. However, limited research examined the association between food/nutrient intake and indexes of sleep in middle-aged and older population in Singapore. Therefore, with a growing number of elderly, studies on improving their sleep quality can play a significant role in improving their quality of life. This is a cross-sectional study and subjects require a 1-day visit (one time visit ONLY). Generally healthy middle-aged and older population will be recruited and after the phone screening and validated subjects will complete the medical history questionnaire and to be brought on the day of visit. During the visit, subjects will stay approximately 3-h to complete the testing. After completing the consent form, fasting-state blood collection and general health assessment will be conducted. Then subjects will be asked to complete the questionnaires to assess sleep quality and dietary intake.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to give an informed consent
2. Age 50 to 75 years
3. Not taking dietary supplements which may impact the outcome of the interests (I.e. dietary protein and vitamin supplements)
4. Not having significant dietary changes for the past 1 year (i.e. weight loss, vegetarian diet)
5. Having sufficient venous access to allow the blood collection
6. Willing to follow the study procedure

Exclusion Criteria:

1. Unable to give an informed consent
2. Age < 50 years
3. Taking dietary supplements which may impact the outcome of the interest (i.e. dietary proteins and vitamin supplements)
4. Having/had significant dietary changes for the past 1 year
5. Not having sufficient venous access to allow the blood collection
6. Unwilling to follow the study procedure

Ages: 50 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study population includes middle-aged and older adults (aged 50 to 75 years) who are in general good health and not regularly having protein or vitamin supplements.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2018-08-02 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jung Eun Kim, PhD, RD, Principal Investigator — NUS (Chemistry, FST)
Locations (1):
- Investigational Medical Unit (IMU), Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Electronic copies of the data with identifiable participant information will be kept on a secure computer with access limited to the principal investigator and her research staff. All data will be de-identified prior to statistical analyses

REFERENCES:
- [Result] Smagula SF, Koh WP, Wang R, Yuan JM. Chronic disease and lifestyle factors associated with change in sleep duration among older adults in the Singapore Chinese Health Study. J Sleep Res. 2016 Feb;25(1):57-61. doi: 10.1111/jsr.12342. PMID 26412328
- [Result] Pan A, De Silva DA, Yuan JM, Koh WP. Sleep duration and risk of stroke mortality among Chinese adults: Singapore Chinese health study. Stroke. 2014 Jun;45(6):1620-5. doi: 10.1161/STROKEAHA.114.005181. Epub 2014 Apr 17. PMID 24743442
- [Result] Dashti HS, Scheer FA, Jacques PF, Lamon-Fava S, Ordovas JM. Short sleep duration and dietary intake: epidemiologic evidence, mechanisms, and health implications. Adv Nutr. 2015 Nov 13;6(6):648-59. doi: 10.3945/an.115.008623. Print 2015 Nov. PMID 26567190
- [Derived] Tan D, Sutanto CN, Lin JWX, Toh DWK, Le KA, Kim JE. Measures of carbohydrate quality and their association with diet quality and cardiometabolic health outcomes in Singapore middle-aged and older adults. Nutr Metab Cardiovasc Dis. 2023 Apr;33(4):778-788. doi: 10.1016/j.numecd.2023.01.008. Epub 2023 Jan 16. PMID 36842956
- [Derived] Toh DWK, Sutanto CN, Loh WW, Lee WY, Yao Y, Ong CN, Kim JE. Skin carotenoids status as a potential surrogate marker for cardiovascular disease risk determination in middle-aged and older adults. Nutr Metab Cardiovasc Dis. 2021 Feb 8;31(2):592-601. doi: 10.1016/j.numecd.2020.10.016. Epub 2020 Oct 26. PMID 33358716

RESULTS

PARTICIPANT FLOW:
Groups:
- Food/Nutrient Intake and Sleep Quality: Cross-sectional research design:
  * fasting-state blood data (plasma amino acids)
  * general health assessment (e.g. blood pressure, anthropometric measurement)
  * dietary data
  * stress and sleep quality assessment
Period: Overall Study
Arm/Group | Food/Nutrient Intake and Sleep Quality
Started | 108
Completed | 108
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Association Between Food/Nutrient Intake and Sleep Quality: This is a cross-sectional study and it does not have an arm/group
Arm/Group | Association Between Food/Nutrient Intake and Sleep Quality
Number analyzed (Participants) | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62
  Male | 46
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Chinese | 94
  Race: Caucasian | 4
  Race: Malaysian | 3
  Race: Indian | 6
  Race: Others | 1

OUTCOME MEASURES:

1. Primary Outcome: Sleep Quality Assessment 1 (GSS)
Description: Pittsburgh sleep quality index (PSQI)
  Global Sleep Score (GSS): 0-21 (arbitrary unit; au) A lower value indicates better sleep quality
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Good Sleep Quality: GSS<=5
- Poor Sleep Quality: GSS>5
- Overall Data: Overall subject data
Arm/Group | Good Sleep Quality | Poor Sleep Quality | Overall Data
Number analyzed (Participants) | 65 | 39 | 104
score on a scale | 3.4 (1.3) | 8.1 (1.9) | 5.2 (2.8)

2. Primary Outcome: Sleep Quality Assessment 2
Description: Sleep evaluation questionnaire
  Score: 0-56 (arbitrary unit) Lower score suggests better sleep
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Good Sleep Quality: GSS=<5
Arm/Group | Good Sleep Quality | Poor Sleep Quality | Overall Data
Number analyzed (Participants) | 65 | 39 | 104
score on a scale | 5.54 (2.32) | 9.08 (3.69) | 6.87 (3.37)

3. Primary Outcome: Dietary Assessment
Description: Food Frequency Questionnaire (FFQ)
Time Frame: Day 1
Reporting Status: Not Posted

4. Primary Outcome: Dietary Assessment 2 (Dietary Carotenoids)
Description: 3 Day 24-Hr Dietary Recall: Participants will be given a diagram showing serving sizes that they can refer to for measurements. Only 3 out of the 7 days of the week are required for the participants to record their food intake. Results are reported as the average value of the analysed nutrients (dietary carotenoids) across the 3 days the dietary data was collected.
Time Frame: Day 3
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Good Sleep Quality | Poor Sleep Quality | Overall Data
Number analyzed (Participants) | 65 | 39 | 104
mg | 11.6 (8.8) | 8.8 (6.7) | 10.5 (8.1)

5. Primary Outcome: Blood Amino Acid Concentration (Plasma Tryptophan)
Description: Amino acid analysis on collected blood serum for blood amino acid profile.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: nmol/mL
Arm/Group | Good Sleep Quality | Poor Sleep Quality | Overall Data
Number analyzed (Participants) | 65 | 39 | 104
nmol/mL | 21.6 (9.2) | 24.7 (11.3) | 22.8 (10.1)

6. Primary Outcome: Dietary Assessment 2 (Dietary Macronutrients)
Description: 3 Day 24-Hr Dietary Recall: Participants will be given a diagram showing serving sizes that they can refer to for measurements. Only 3 out of the 7 days of the week are required for the participants to record their food intake. Results are reported as the average value of the analysed nutrients (dietary fat) across the 3 days the dietary data was collected.
Time Frame: Day 3
Measure: Mean (Standard Deviation); unit: percentage of energy intake
Arm/Group | Good Sleep Quality | Poor Sleep Quality | Overall Data
Number analyzed (Participants) | 65 | 39 | 104
percentage of energy intake
  Total Fat | 34.3 (6.4) | 32.8 (7) | 33.7 (6.6)
  Total Carbohydrate | 47.3 (6.8) | 48.1 (8.7) | 47.6 (7.5)
  Total Protein | 18.4 (4.0) | 19.1 (4.2) | 18.7 (4.1)

7. Primary Outcome: Sleep Quality Assessment 1 (Sleep Duration)
Description: Pittsburgh sleep quality index (PSQI)
  Sleep duration (hours)
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Good Sleep Quality | Poor Sleep Quality | Overall Data
Number analyzed (Participants) | 65 | 39 | 104
hours | 6.7 (1.1) | 6.2 (1.3) | 6.5 (1.2)

8. Primary Outcome: Sleep Quality Assessment 1 (Sleep Latency)
Description: Pittsburgh sleep quality index (PSQI)
  Sleep latency (minutes)
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Good Sleep Quality | Poor Sleep Quality | Overall Data
Number analyzed (Participants) | 65 | 39 | 104
minutes | 10 (7.6) | 26 (17.7) | 16.0 (14.5)

9. Primary Outcome: Sleep Quality Assessment 1 (Sleep Efficiency)
Description: Pittsburgh sleep quality index (PSQI)
  Sleep efficiency (%)
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: percentage of sleep from time in bed
Arm/Group | Good Sleep Quality | Poor Sleep Quality | Overall Data
Number analyzed (Participants) | 65 | 39 | 104
percentage of sleep from time in bed | 93.9 (5.8) | 84.6 (9.7) | 90.4 (8.7)

10. Secondary Outcome: Blood Pressure
Description: Blood pressure using electronic devices that work on the oscillometric technique. The systolic and diastolic blood pressure are both collected and reported
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Good Sleep Quality | Poor Sleep Quality | Overall Data
Number analyzed (Participants) | 65 | 39 | 104
mmHg
  Systolic Blood Pressure | 118.9 (16.1) | 113.4 (18.4) | 116.8 (17.1)
  Diastolic Blood Pressure | 76 (10.2) | 73.1 (11.3) | 74.9 (10.7)

11. Secondary Outcome: Anthropometric Measurements 1
Description: Height (kg)
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Good Sleep Quality | Poor Sleep Quality | Overall Data
Number analyzed (Participants) | 65 | 39 | 104
cm | 161.9 (7.9) | 160.2 (8.9) | 161.3 (8.3)

12. Secondary Outcome: Anthropometric Measurements 2
Description: Weight (kg)
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Good Sleep Quality | Poor Sleep Quality | Overall Data
Number analyzed (Participants) | 65 | 39 | 104
kg | 63.2 (14.0) | 60.7 (11.6) | 62.3 (13.1)

13. Secondary Outcome: Anthropometric Measurements 3
Description: Waist circumference (cm)
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Good Sleep Quality | Poor Sleep Quality | Overall Data
Number analyzed (Participants) | 65 | 39 | 104
cm | 83.6 (13.1) | 81.5 (10.3) | 82.8 (12.1)

14. Secondary Outcome: Skin Carotenoid Status
Description: Measure with resonance Raman spectroscopy. A higher score is indicative of raised skin carotenoid levels and hence, a better outcome
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Good Sleep Quality | Poor Sleep Quality | Overall Data
Number analyzed (Participants) | 65 | 39 | 104
score on a scale | 32746 (11195) | 35307 (13139) | 33707 (11963)

15. Secondary Outcome: Perceived Stress Assessment
Description: Perceived stress assessment (PSS) questionnaire
  Score: 0-40 (arbitrary unit; au) A higher score indicates higher perceived stress
Time Frame: Day 1
Population: Current data is the overall mean of the subjects that has participated. Comparison analysis is incomplete and still in progress.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Good Sleep Quality | Poor Sleep Quality | Overall Data
Number analyzed (Participants) | 65 | 39 | 104
score on a scale | 10.5 (5.3) | 14.8 (5.8) | 12.1 (5.8)

16. Secondary Outcome: Blood Lipid and Glucose Profile
Description: Plasma triglycerides, total cholesterol, ldl-cholesterol, hdl-cholesterol and glucose concentration
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Good Sleep Quality | Poor Sleep Quality | Overall Data
Number analyzed (Participants) | 65 | 39 | 104
mmol/L
  Triglyceride | 1.23 (0.57) | 1.16 (0.54) | 1.20 (0.56)
  Total cholesterol | 5.4 (1.0) | 5.3 (1.0) | 5.3 (1.0)
  LDL-cholesterol | 3.22 (0.88) | 3.15 (0.94) | 3.19 (0.90)
  HDL-cholesterol | 1.58 (0.48) | 1.62 (0.45) | 1.60 (0.47)
  Glucose | 5.50 (0.89) | 5.37 (1.26) | 5.5 (1.0)

17. Secondary Outcome: Plasma Carotenoids Concentration
Description: High performance liquid chromatography quantitative analyses of carotenoids in plasma samples
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Good Sleep Quality | Poor Sleep Quality | Overall Data
Number analyzed (Participants) | 65 | 39 | 104
mg/L | 1.14 (0.51) | 1.22 (0.76) | 1.17 (0.61)

ADVERSE EVENTS:
Time Frame: 1 Year.
Description: Definition is the same as clinicaltrials.gov
Arm/Group | Association Between Food/Nutrient Intake and Sleep Quality
All-Cause Mortality (participants affected / at risk) | 0/108
Serious Adverse Events (participants affected / at risk) | 0/108
Other Adverse Events (participants affected / at risk) | 0/108

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2019-10-31): https://cdn.clinicaltrials.gov/large-docs/54/NCT03554954/Prot_ICF_000.pdf